CLINICAL TRIAL: NCT04605211
Title: Being Present-MPN: A Distress Reduction Intervention for Patients With BCR-ABL-Negative MPNs and CML on Tyrosine Kinase Inhibitors
Brief Title: A Distress Reduction Intervention for Patients With BCR-ABL-Negative MPNs or CML on Tyrosine Kinase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202510; NCI-2020-07364 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Myeloproliferative Neoplasm; Chronic Phase Chronic Myelogenous Leukemia; Chronic Myeloid Leukemia
Keywords: BCR-ABL-Negative; Distress Reduction; Tyrosine Kinase Inhibitors; Leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Being Present (Supportive Care) (Experimental): Patients and caregivers receive Being Present intervention consisting of online audio-based mindfulness meditation exercise over 15 minutes at least 5 times per week, daily meditation reminders, and online webinars over 30-60 minutes every week.
  Interventions: Behavioral: Online Mindfulness Meditation; Other: Internet-Based Webinars

INTERVENTIONS:
Behavioral: Online Mindfulness Meditation — Complete online audio-based mindfulness meditation exercises
  Other Names: Online MBSR; Online Mindful Meditation; Web-Based Mindfulness Meditation
Other: Internet-Based Webinars — Attend webinars

SUMMARY:
This trial looks at how well a distress reduction intervention, called "Being Present", works to improve the quality of life of patients with BCR-ABL-negative myeloproliferative neoplasms (MPNs) or chronic phase chronic myeloid leukemia (CP-CML) who are taking tyrosine kinase inhibitors (TKIs) and their caregivers. Mindfulness meditation is the practice of repeatedly bringing attention back to the immediate experience and may help people cope with various types of illness, stress, and worry. This may help patients and caregivers to gradually learn to disconnect from reacting to and dwelling on the past and future and instead fully experiencing the present moment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To tailor the Being Present intervention to BCR-ABL-negative MPN and CP-CML patients.

II. To determine the feasibility of an 8-week web-based mindfulness meditation program with live webinars among BCR-ABL-negative MPN patients and their caregivers, and CP-CML patients on tyrosine kinase inhibitors (TKIs), and CP-CML patients in treatment-free remission (TFR).

III. To determine the acceptability of an 8-week web-based mindfulness meditation program with live webinars among BCR-ABL-negative MPN patients and their caregivers, CP-CML patients on TKIs, CP-CML patients on TKIs, and CP-CML patients in TFR.

SECONDARY OBJECTIVE:

I. To evaluate the preliminary efficacy of the intervention.

EXPLORATORY OBJECTIVES:

I. To evaluate for differences in the feasibility and acceptability of an 8-week web-based mindfulness meditation program with live webinars:

Ia. Based on demographic or clinicopathologic factors. Ib. In patients versus caregivers.

II. To evaluate for differences in the preliminary efficacy an 8-week web-based mindfulness meditation program with live webinars:

IIa. Based on demographic or clinicopathologic factors. IIb. In BCR-ABL-negative patients versus caregivers. IIc. In BCR-ABL-negative patient-caregiver pairs versus unpaired patients. IId. Based on level of adherence to the practice instructions.

OUTLINE:

Patients and caregivers receive Being Present intervention consisting of online audio-based mindfulness meditation exercise over 15 minutes at least 5 times per week, daily meditation reminders, and online webinars over 30-60 minutes every week.

After completion of study, patients and caregivers are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Carry a diagnosis of BCR-ABL-negative MPN or CML
* PATIENT: Have an estimated life expectancy of at least 6 months, assessed by principal investigator or treating investigator
* PATIENT: Be able to speak and read English
* PATIENT: Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet (assessed by participant self-report)
* PATIENT: Have daily access to a mobile phone capable of receiving text messages, as determined by a study investigator
* PATIENT: Be able to provide informed consent
* CAREGIVER: Be a spouse/partner, other family member, or a close friend of a BCR-ABL-negative patient who consented to participate in the Being Present-MPN study
* CAREGIVER: Be able to speak and read English
* CAREGIVER: Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet (assessed by participant self-report)
* CAREGIVER: Have access to a mobile phone capable of receiving text messages, as determined by a study investigator
* CAREGIVER: Be able to provide informed consent

Exclusion Criteria:

* PATIENT: Have had their BCR-ABL-negative MPN transform into acute leukemia
* PATIENT: Have had their CP-CML transform into blast phase
* PATIENT: Be post-allogeneic stem cell transplantation
* PATIENT AND CAREGIVER: Have extensive hearing loss such that ability to participate in the study would be impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Primary Symptoms | Up to 90 days
  The frequency of primary symptoms will be categorized and assessed by semi-structured qualitative interviews.
Frequency of Participants' Understanding of Hematologic Malignancies | Up to 90 days
  The frequency and categorization of participants' understanding of hematologic malignancies will be assessed by semi-structured qualitative interviews.
Frequency of Participants' Perception of web-based mindfulness meditation | Up to 90 days
  The frequency and categorization of participants' perception of web-based mediation will be assessed by semi-structured qualitative interviews.
Frequency of Reported Barriers of Web-Based Mindfulness Meditation | Up to 90 days
  The frequency and categorization of participants' reported barriers to web-based mediation will be assessed by semi-structured qualitative interviews.
Percentage of patients approached who consent to participate | Up to 90 days
  Recruitment rate will be reported as a percentage of all patients who were approached by the study team or medical professional whom consented to participate in the active study.
Frequency of Reasons for Ineligibility | Up to 90 days
  For potential study candidates who are ineligible, caregiver relationship and reasons for ineligibility will be collected. Reasons for ineligibility will be reported using descriptive statistics.
Frequency of Reasons for Refusal to Participate | Up to 16 weeks
  For potential study candidates who decide not to participate, caregiver relationship and reasons for refusal will be collected. Reasons for refusal will be reported using descriptive statistics.
Frequency of Attrition over time | Up to 16 weeks
  The number of participants who attend the web-based sessions will be recorded via a roll-call and recorded at each study visit.
Frequency of Attrition Causes | Up to 16 weeks
  Reasons for not attending the web-based interventions will be recorded and characterized. Reasons for attrition will be reported using descriptive statistics.
Frequency of meditation practice | Up to 16 weeks
  The study team will call participants and conduct a brief interview to gauge current mindfulness meditation practice. Frequency of mediation will be reported using descriptive statistics.
Median duration of meditation practice | Up to 16 weeks
  The study team will call participants and conduct a brief interview to gauge current duration of mindfulness meditation practice. Duration of mediation will be reported using descriptive statistics.
Frequency of playing recorded webinars | Up to 16 weeks
  The frequency in which participants utilize the recorded webinars will be captured via website data and will be reported using descriptive statistics
Duration of playing recorded webinars | Up to 16 weeks
  The duration in which participants utilize the recorded webinars will be captured via website data and will be reported using descriptive statistics
Measure of Acceptability using semi-structured interviews | Up to 16 weeks
  Information about acceptability and the overall intervention experience will come from semi-structured interviews. Audio recordings of the semi-structured interviews will be professionally transcribed and coded using Atlas.ti for categorizing acceptability using qualitative thematic analysis by at least two investigators.

SECONDARY OUTCOMES:
Mean change in scores on the National Comprehensive Cancer Network (NCCN) Distress Thermometer scores | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  This single-item inventory uses an analog graphic to allow patients to assess their overall distress with a score range of 0 (no distress) to 10 (extreme distress). A score of 4 or higher to differentiate clinically significant distress. Paired t-tests will compare validated survey results.
Mean change in scores on the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The PROMIS anxiety scale is a 8 item scale which measures a participants anxiety based on their response to anxiety related items. Each item response ranges from 1 (never) to 5 (always)Paired t-tests will compare validated survey results. Raw scores ranging from 8 - 40 are converted to scaled scores to determine a standardized anxiety score with higher scores indicating a greater anxiety. Paired t-tests will compare validated survey results.
Mean change in scores on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The EORTC QLQ-C30 has been developed as a quantitative measure of health-related quality of life for use in clinical trials of cancer patients. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. Paired t-tests will compare validated survey results.
Mean change in scores on the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The MPN-SAF TSS is 10-item questionnaire is recommended in the NCCN Guidelines for the assessment of symptom burden at baseline and monitoring symptom status during the course of treatment with individual item scores ranging from 0 (absent) to 10 (worst imaginable). Total Scores range from 0-100, with higher scores indicating a greater number of symptoms and severity. Paired t-tests will compare validated survey results.
Mean change in scores on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-CML24) | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The EORTC QLQ-CML24 assessment consists of 24 items measuring the following aspects: Symptom Burden, Impact on Daily Life, Impact on Worry/Mood, Body Image Problems, Satisfaction with Care and Satisfaction with Social Life. This scale includes 24 items with responses ranging from a score of 0 (not at all) to 4 (very much). Paired t-tests will compare validated survey results.
Mean change in scores on the Caregiver Quality of Life Index - Cancer (CQOLC) | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The CQOLC is a self-administered scale specifically designed to evaluate cancer patient caregiver quality of life. This scale includes 35 items with responses ranging from a score of 0 (not at all) to 4 (very much). The total possible score is 140, with higher scores representing better quality of life. Paired t-tests will compare validated survey results.
Mean change in scores on the Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | Baseline, 4 weeks, and 8 weeks, Up to 8 weeks total
  The FFMQ-SF assessment measures five facets of mindfulness: Observing, Describing, Acting with Awareness, Non-Judging of inner experience, and Non-Reactivity to inner experience. The score of each facet is computed by summing the 3 items assigned to the facet which asks the individual to rate which response represents your own opinion of what is generally true for you. Each statement (item) has scores ranging from 1 (never or very rarely true) to 5 (very often or always true), for a total of 15 points per facet. Paired t-tests will compare validated survey results.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Schoenbeck, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No